CLINICAL TRIAL: NCT03389373
Title: Microbial Testing for Caries Risk Assessment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Saliva testing was not sensitive enough to correctly identify high risk patients
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-1535
Record Dates: First submitted 2017-12-22; First posted 2018-01-03 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Dental Caries
Keywords: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Children will have a saliva sample analyzed for amount of bacteria. Children who have higher bacteria counts are at higher risk of developing cavities.
Masking Description: Provider and investigator will know if child has clinical caries or not at the time of saliva sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Child with full primary dentition (Other): All children who match inclusion criteria are eligible to have a saliva sample obtained which will act as a proxy for bacterial levels. High bacteria levels are correlated with a higher risk of developing cavities.
  Interventions: Device: GC Strep Mutans Saliva Sampling

INTERVENTIONS:
Device: GC Strep Mutans Saliva Sampling — Children who match inclusion criteria will have a saliva sample obtained which will act as a proxy for bacterial levels.

SUMMARY:
Specific Aims

1) Assess CG (Cariogenic) Saliva-Check Mutans® saliva testing for identification of high caries risk patients

DETAILED DESCRIPTION:
Hypotheses and Specific Aims

Hypotheses CG Saliva-Check Mutans will test positive in children with clinical caries.

Specific Aims

* Assess CG Saliva-Check Mutans saliva testing for identification of high caries risk patients

Background and Significance

Early Childhood Caries

Suboptimal oral health is an existing and growing concern for the pediatric patient, with dental decay considered the most common chronic disease of childhood in the United States. About 1 in 5 children (20%) aged 5 to 11 years old have at least one untreated decayed tooth, with childhood caries being 4 times more common than early childhood obesity, 5 times more common than asthma, and 20 times more common than diabetes. Early childhood caries (ECC) is diagnosed when one or more primary teeth are affected by the caries process before six years of age, and severe early childhood caries (S-ECC) is defined as any smooth-surface caries in a child under the age of three. ECC is a multifactorial process and is not exclusively associated with poor feeding habits such as ad libitum bottle or breast-feeding. Factors include susceptible tooth surfaces, frequent consumption of a cariogenic diet, and an elevated colonization of cariogenic bacteria. Mutans Streptococci (MS) are pathognomonic for ECC and S-ECC in all age groups. The rise of ECC and S-ECC has increased the number of children needing dental treatment at an early age, often requiring treatment in advanced care settings such as under sedation, general anesthesia, or the emergency department. Over 51 million school hours are lost each year due to dental problems or urgent dental needs. Furthermore, 44 % of children in the U.S. will suffer from pediatric dental disease before kindergarten and approximately 22% of people across all age groups have existing untreated dental decay. As health care providers, it is imperative for both dentists and pediatricians to promote optimal oral health through the utilization of prevention strategies, such as the caries risk assessment.

Caries Risk Assessment (CAMBRA)

The multiple factors that contribute to dental caries development should be evaluated to determine an individual patient's risk status. An evidence-based model termed Caries Management Risk Assessment (CAMBRA) was developed to provide dentists with a protocol for caries diagnosis, prevention and treatment. CAMBRA helps identify children at risk of caries development and provides age-specific recommendations for caries prevention across all demographics. The goal of the assessment is that by identifying a patient at high risk of caries development, the dental provider can make patient specific recommendations in attempt to lower risk and mitigate disease progression. The risk assessment for all patients determines biological, protective, and clinical factors that may contribute to the caries disease process. Examples of high risk factors for pediatric patients include frequent between meal sugar-containing foods and sugar sweetened beverages (SSB), nighttime bottle feeding, previous caries experience, and elevated MS levels. Protective factors against caries progression include optimal oral hygiene, topical fluoride, and sugar substitutes.

Concepts of a Healthy Mouth

A healthy mouth has a symbiotic environment of cariogenic and non-cariogenic bacteria and is characterized as being free of and at low risk for developing disease. A low plaque score (or low plaque growth) has a strong correlation with a healthier mouth for both dental and periodontal health. When the symbiotic relationship becomes unbalanced, the resulting acidic environment leads to demineralization of tooth structure. High levels of cariogenic bacteria such as Mutans Streptococci (MS) and Lactobacilli acidophilus (LB) lower environmental pH levels, which selects for progressive dissolution of mineral into saliva and causes an increased risk of caries development. Saliva is an important intrinsic host factor protecting against caries formation, as it provides a reservoir of calcium, phosphate and fluoride to remineralize affected enamel and acts as a buffer to reestablish a healthy oral pH. By educating parents of the pediatric patient about concepts of a healthy mouth and demonstrating good oral hygiene practices, a child can be at lower risk for dental decay.

Etiology of Caries

Dental caries is a multifactorial disease process that is driven primarily by a diet high in fermentable carbohydrates and simple sugars, cariogenic bacteria, and suboptimal oral hygiene. The prevailing microorganisms that contribute to the development of dental caries are MS and LB, which metabolize fermentable carbohydrates to produce acid (acidogenic) and thrive in low pH environments (aciduric). Frequent consumption of fermentable carbohydrates and SSBs leads to maintained levels of low salivary pH, resulting in the dissolution of calcium and phosphate from enamel surfaces over time. This demineralization of tooth structure presents initially as a white spot lesion, which can be reversed or remineralized by decreasing exposure to fermentable carbohydrates and practicing optimal oral hygiene. However, if the local oral environment is not improved to promote remineralization at these affected sites, mineral loss will continue until a physical breakdown or cavitation of the enamel's crystal lattice structure occurs, requiring surgical intervention to restore.

Prevention Measures and Adjective Therapies (Prevident5000)

Fluoride applications represent a non-surgical approach to enamel remineralization. High concentrations of fluoride, such as those found in toothpastes and varnishes, creates an altered layer of calcium (fluorapatite) on the tooth surface. Therefore, fluoride aides to increase the pH for acid resistance and decrease the adhesion of bacteria to smooth surfaces by directly affecting the metabolism activity of cariogenic bacteria. High fluoride containing toothpastes such as PreviDent5000 Plus (1.1 % NaF; 5,000ppm F) has been shown to be effective at increasing enamel remineralization and reducing dental caries in both the primary and permanent dentition. When used as an at home regimen, PreviDent5000 decreased lesion depths up to 24%, supporting the finding that dentifrices with 5,000ppm fluoride are more effective at remineralizing carious lesions compared to standard over the counter dentifrices containing 1,100 - 1,500ppm fluoride. However, it remains unclear if PreviDent5000 Plus has been effective in decreasing caries causing bacteria.

Background on Salivary Testing Various salivary tests have been used for years in clinical practice to determine a patient's oral bacterial load. Culturing MS from saliva in children has proven safe and valuable as part of a caries risk assessment due to the correlation between high bacterial levels and caries development. Saliva testing is relatively simple with a previous study completed at the Children's Hospital Colorado Pediatric Dentistry Clinic supporting the efficacy of several different methods for saliva collection, including directly pipetting saliva, swabbing the buccal surfaces of teeth, and stimulating saliva production with a paraffin pellet. Saliva is obtained and cultured for bacteria that are causative in caries initiation and progression, such as MS and LB. Children with a high load of MS have been shown to be 6 times more likely to develop caries and experience caries progress over a five-year period. GC Saliva-Check Mutans has been used in dental practices as a useful and simple microbial testing tool to aide providers in caries risk detection. Bacterial (MS) samples resulting in 5x10 to the 5th power colony-forming units per milliliter of saliva (CFU/mL) indicates a low caries risk. In contrast, less than 5x10 to the 5th power CFU/mL of MS in a saliva sample correlates to a moderate or high caries risk. This study is designed to use saliva sampling to determine a non-surgical adjunctive therapy to help lower cavity causing bacteria. The value of saliva testing is that it can serve as both a non-invasive diagnostic tool in determining a patient's caries risk status and a visual aide for educating parents and young patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be a patient of record at Children's Hospital Colorado Dental Center
* Child must fall between 24 and 96 months of age
* Child must present with full primary dentition

Exclusion Criteria:

* Patients with a complex medical history classified as being greater than ASA II
* Patients with recent dose of antibiotics within the previous two weeks or who present with a low caries risk set forth by the AAPD

Ages: 24 Months to 96 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Count of Strep Mutans bacterial | 4 weeks
  Bacterial (MS) samples resulting in〖5x10〗^5 colony-forming units per milliliter of saliva (CFU/mL) indicates a low caries risk. In contrast, >〖5x10〗^5 CFU/mL of MS in a saliva sample correlates to a moderate or high caries risk. This study is designed to use saliva sampling to determine a non-surgical adjunctive therapy to help lower cavity causing bacteria.

SECONDARY OUTCOMES:
Plaque Index | 4 weeks
  An index for estimating the status of oral hygiene by measuring dental plaque that occurs in the areas adjacent to the gingival margin. A score of 0 to 3 (0=no plaque, 1=minimal plaque, 2 = moderate plaque, 3= extensive plaque is assigned to each of 5 division on the tooth). The score is then divided by 5. The patient's resultant plaque rating is considered excellent if the score is 0, Good if it is between 0.1-1.7, Fair if it is between 1.8-3.4 and Poor if it is between 3.5-5. The hope is to see a reduction of plaque score in study participants at the follow-up visit 4 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Camille V Gannam, DMD MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children'S Hospital Colorado Dental Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
This is a small resident research project comparing the effect of Prevident5000 plus versus over the counter toothpaste on cariogenic bacteria counts as well as the effect of frequent hygiene reminders on oral hygiene (plaque score).

REFERENCES:
- [Result] Dye BA, Li X, Beltran-Aguilar ED. Selected oral health indicators in the United States, 2005-2008. NCHS Data Brief. 2012 May;(96):1-8. PMID 23050519
- [Result] Larson K, Cull WL, Racine AD, Olson LM. Trends in Access to Health Care Services for US Children: 2000-2014. Pediatrics. 2016 Dec;138(6):e20162176. doi: 10.1542/peds.2016-2176. Epub 2016 Nov 15. PMID 27940710
- [Result] Mills C, Patel P. Adopting caries risk assessment in all practice environments. Gen Dent. 2016 Jul-Aug;64(4):66-72. PMID 27367637
- [Result] Edelstein BL, Ureles SD, Smaldone A. Very High Salivary Streptococcus Mutans Predicts Caries Progression in Young Children. Pediatr Dent. 2016;38(4):325-30. PMID 27557922
- [Result] Li Y, Argimon S, Schon CN, Saraithong P, Caufield PW. Characterizing Diversity of Lactobacilli Associated with Severe Early Childhood Caries: A Study Protocol. Adv Microbiol. 2015 Jan 1;5(1):9-20. doi: 10.4236/aim.2015.51002. PMID 26413427
- [Result] Leone CW, Oppenheim FG. Physical and chemical aspects of saliva as indicators of risk for dental caries in humans. J Dent Educ. 2001 Oct;65(10):1054-62. PMID 11699977
- [Result] Thibodeau EA, O'Sullivan DM, Tinanoff N. Mutans streptococci and caries prevalence in preschool children. Community Dent Oral Epidemiol. 1993 Oct;21(5):288-91. doi: 10.1111/j.1600-0528.1993.tb00776.x. PMID 8222603
- [Result] Lee C, Tinanoff N, Minah G, Romberg E. Effect of Mutans streptococcal colonization on plaque formation and regrowth in young children--a brief commnunication. J Public Health Dent. 2008 Winter;68(1):57-60. doi: 10.1111/j.1752-7325.2007.00050.x. PMID 18494159
- [Result] Amaechi BT, Ramalingam K, Mensinkai PK, Chedjieu I. In situ remineralization of early caries by a new high-fluoride dentifrice. Gen Dent. 2012 Jul-Aug;60(4):e186-92. PMID 22782050
- See also: Guideline on Fluoride Therapy — http://www.aapd.org/media/policies_guidelines/g_fluoridetherapy.pdf
- See also: Guideline on Caries-risk Assessment and Management for Infants, Children, and Adolescence — http://www.aapd.org/media/policies_guidelines/g_cariesriskassessment.pdf
- See also: Policy on Early Childhood Caries (ECC): Unique Challenges and Treatment Options — http://www.aapd.org/media/policies_guidelines/p_eccclassifications.pdf